CLINICAL TRIAL: NCT03642704
Title: HIV Diagnosis and Treatment at Birth for HIV Exposed Newborn Whose Mother Was Not Treated With Antiretroviral Therapy (ART) During Last Month Before Delivery : Strategy Evaluation in Guinea.
Brief Title: HIV Diagnosis and Treatment at Birth for Newborn With High Risk HIV Exposure
Acronym: DIAVINA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS12344-DIAVINA
Record Dates: First submitted 2017-03-20; First posted 2018-08-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Mother to Child HIV Transmission
Keywords: PMTCT; HIV early diagnosis; HIV preventive therapy; prevention of mother to child HIV transmission

STUDY DESIGN:
Intervention Model Description: Prospective non-comparative study of mother-child pairs whose mother is HIV-infected and received less than 4 weeks of antiretroviral therapy before birth or whose HIV infection has been diagnosed at birth. Assess the operational efficacy of a strategy combining early diagnosis and preventive antiretroviral treatment systematically reinforced from the birth among infants at high risk of infection with HIV.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reinforced preventive ARV therapy (Experimental): The proposed reinforced preventive ARV Therapy will be administrated to all newborns exposed to HIV (zidovudine+lamivudine+nevirapine if the newborn is exposed to HIV-1 or HIV-1/2, zidovudine+lamivudine if the newborns exposed to HIV-2)
  Interventions: Drug: Reinforced preventive ARV therapy

INTERVENTIONS:
Drug: Reinforced preventive ARV therapy — If the mother is HIV-1 or HIV 1/2 infected:
  * zidovudine / laminvudine (60/30 mg), ¼ cp morning and evening orally for 12 weeks.
  * nevirapine: 15mg/OD if weight ≥ 2500g / 10mg/OD if weight = 2000-2499g / 2mg/kg/OD if weight < 2000g for 12 weeks in case of HIV-1 infection. After 6 weeks, nevirapine will increase at 20mg/OD
  If the mother is HIV-2 infected:
  - zidovudine / laminvudine (60/30 mg), ¼ cp morning and evening orally for 12 weeks.
  Other Names: Early diagnosis in children exposed to HIV

SUMMARY:
Principal objective Assess the operational efficacy of a strategy combining early diagnosis and preventive antiretroviral treatment systematically reinforced from the birth* among infants at high risk of infection with HIV** .

* in a maximum of 48 hours after delivery

  * born from HIV infected mothers who received less than 4 weeks of antiretroviral therapy prior delivery and / or HIV infection diagnosed at delivery

Intervention, a combined strategy :

After positive HIV infection screening from mother in the delivery room and put on antiretroviral treatment of mothers with post partum according to national guidelines , newborns benefit :

* Early detection of HIV infection at birth
* Without awaiting the outcome of early detection result, a preventive reinforced antiretroviral treatment (zidovudine, lamivudine, nevirapine or zidovudine, lamivudine if their mother is infected with HIV-2), from birth for 12 weeks.
* Regular HIV screening until the end of breastfeeding or later to 18 months.
* In case of positive results of an HIV test, an antiretroviral treatment with zidovudine, lamivudine, lopinavir, ritonavir whatever serology HIV 1 or 2.

DETAILED DESCRIPTION:
Objectives Principal objective Assess the operational efficacy of a strategy combining early diagnosis and preventive antiretroviral treatment systematically reinforced from the birth* among infants at high risk of infection with HIV** .

* in a maximum of 48 hours after delivery

**born from HIV infected mothers who received less than 4 weeks of antiretroviral therapy prior delivery and / or HIV infection diagnosed at delivery Secondary objectives

* Measure the cascade management of HIV infected mothers and HIV infected infants
* Measure the tolerance of reinforced preventive antiretroviral treatment
* Describe the rate of mother to child transmission of HIV and its risk factors
* Describe the clinical and immuno-virologic outcomes in mothers, in HIV infected children and in HIV-non-infected children
* Evaluate the acceptability of the strategy by mothers and caregivers.
* Compare the early diagnosis of HIV infection with Abbott and Biocentric HIV RNA tests

Methodology Prospective non-comparative study of mother-child pairs whose mother is HIV-infected and received less than 4 weeks of antiretroviral therapy before birth or whose HIV infection has been diagnosed at birth.

Estimated enrolment: 300 mother-child pairs

Eligibility:

Inclusion criteria:

Mother-child pairs whose mother is HIV-infected and received less than 4 weeks of antiretroviral therapy before delivery or whose HIV infection has been diagnosed at delivery Mother who signed the informed consent form to participate in the study.

non-inclusion criteria: Mother treated with antiretrovirals during the month preceding delivery No inclusion for precautionary reason : clinical symptoms suggesting an opportunistic infection of the central nervous system.

No inclusion for monitoring difficulties History or presence of allergy to the study drugs or their components Contra-indications to the study drugs Symptoms, physical signs or laboratory values suggestive of systemic disorders, (including renal, hepatic, cardiovascular, pulmonary, skin, or psychiatric and other conditions, which could interfere with the interpretation of the trial results

Intervention, a combined strategy :

After positive HIV infection screening from mother in the delivery room and put on antiretroviral treatment of mothers with post partum according to national guidelines , newborns benefit :

* Early detection of HIV infection at birth
* Without awaiting the outcome of early detection result, a preventive reinforced antiretroviral treatment (AZT / 3TC / NVP or AZT / 3TC if their mother is infected with HIV -2), from birth for 12 weeks.
* Regular HIV screening until the end of breastfeeding or later to 18 months.
* In case of positive results of an HIV test, an antiretroviral treatment with AZT / 3TC / LPV whatever serology HIV 1 or 2.

ELIGIBILITY:
Inclusion Criteria:

* Mother-child pairs whose mother is HIV-infected and received less than 4 weeks of antiretroviral therapy before delivery or whose HIV infection has been diagnosed at delivery
* Mother who signed the informed consent form to participate in the study.

Exclusion Criteria:

* Mother treated with antiretrovirals during the month preceding delivery
* No inclusion for precautionary reason : clinical symptoms suggesting an opportunistic infection of the central nervous system.
* No inclusion for monitoring difficulties
* History or presence of allergy to the study drugs or their components
* Symptoms, physical signs or laboratory values suggestive of systemic disorders, (including renal, hepatic, cardiovascular, pulmonary, skin, or psychiatric and other conditions, which could interfere with the interpretation of the trial results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Proportion of newborns who have received an HIV diagnosis and reinforced preventive antiretroviral treatment at birth. | Day 2
  Proportion of newborns who have received both HIV test and reinforced preventive antiretroviral treatment in a maximum of 48 hours after birth.

SECONDARY OUTCOMES:
Proportion of mothers diagnosed with HIV who will initiate an antiretroviral therapy | Week 72
  • Proportion of mothers diagnosed with HIV at Day 0 who will initiate an antiretroviral therapy
Proportion of children diagnosed with HIV who will initiate an antiretroviral therapy | Week 72
  • Proportion of children diagnosed with HIV from Day 0 to Week 72 who will initiate an antiretroviral therapy
Proportion of mother-child pairs retained in the study with child having 2 PCR performed after stopping reinforced preventive antiretroviral treatment | Week 24
  • Proportion of mother-child pairs retained in the study from Day 0 to Week 24 with child having 2 PCR performed after stopping reinforced preventive antiretroviral treatment
Proportion of mother-child pairs retained in the study | Week 72
  • Proportion of mother-child pairs retained in the study from Day 0 to Week 72.

OTHER OUTCOMES:
Measure the clinical tolerance of reinforced preventive antiretroviral treatment in children | Week 12
  • Nature of clinical adverse events
Measure the biological tolerance of reinforced preventive antiretroviral treatment in children | Week 12
  • Nature of biological adverse events
Measure the proportion of children on reinforced preventive antiretroviral treatment with anemia | Week 12
  • Proportion of children with anemia superior or equal to grade 2
Measure the proportion of children who change antiretroviral therapy for grade 4 adverse event | Week 12
  • Proportion of children who change antiretroviral therapy for grade 4 adverse event
Measure the proportion of children with preventive antiretroviral treatment interruption | Week 12
  • Proportion of children with preventive antiretroviral treatment interruption
Describe the clinical events occurring in mothers | Week 72
  • Description of clinical events occurring in mothers
Measure the proportion of mothers presenting clinical events | Week 72
  • Proportion of mothers presenting clinical events
Describe the immunological outcomes in mothers | Week 72
  • Value of CD4 (absolute number)
Describe the virological outcomes in mothers | Week 72
  • Value of HIV RNA (copies/mL)
Describe the clinical outcomes in HIV-infected children | Week 48
  • Description of clinical events occurring in HIV-infected children
Measure the proportion of HIV-infected children presenting clinical events | Week 48
  • Proportion of HIV-infected children presenting clinical events
Describe the immunological outcomes in HIV infected children | Week 48
  • Value of CD4 (absolute number)
Describe the virological outcomes in HIV infected children | Week 48
  • Value of HIV RNA (copies/mL)
Describe the clinical outcomes in HIV-non-infected children | Week 72
  Nature of clinical events occurring in HIV-non-infected children
Measure the proportion of HIV-non-infected children presenting clinical events | Week 72
  • Proportion of HIV-non-infected children presenting clinical events
Describe the rate of mother to child transmission of HIV | Week 72
  • Proportion of HIV infected children (based on PCR ADN or ARN)
Describe the risk factors of mother to child transmission of HIV | week 72
  Description of risk factors for HIV transmission

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Breton, MD, Principal Investigator — Solthis; Mohamed Cisse, MD, Principal Investigator — CHU Donka
Locations (1):
- Hôpital National Ignace Deen, Conakry, Guinea

IPD SHARING:
Plan to Share IPD: No